CLINICAL TRIAL: NCT02127892
Title: Phase I/II Trial of Hematopoietic Stem Cell Transplant (HSCT) for Children With Severe Combined Immune Deficiency (SCID) and Without an HLA-Matched Sibling Donor
Brief Title: SCID Bu/Flu/ATG Study With T Cell Depletion
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed due to slow accrual. Nine subjects enrolled over 7 years.
Sponsor: Neena Kapoor, M.D. (Other)
Responsible Party: Sponsor-Investigator, Neena Kapoor, M.D., Professor of Pediatrics, Keck School of Medicine; Division Head, Division of Research Immunology/BMT, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-06-00243
Record Dates: First submitted 2012-10-19; First posted 2014-05-01 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-08

CONDITIONS: Severe Combined Immunodeficiency
Keywords: Severe Combined Immune Deficiency; SCID; HLA-matched unrelated donor; unrelated; MUD; bone marrow; cord blood; haplo-identical; peripheral blood; CD34+ selection; T cell depletion; HSCT; BMT; CliniMACS
MeSH Terms: conditions — Severe Combined Immunodeficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- unrelated BM with T cell depletion (Other): Acceptable matching for matched unrelated donor (MUD) bone marrow will be genotypic matches at 10 of 10 HLA alleles (HLA-A, B, C, DR and DQ) or 9 of 10 HLA alleles.
  Interventions: Biological: unrelated BM with T cell depletion
- unrelated cord blood (Other): Acceptable matching for unrelated cord blood will be a genotypic match at 6 of 6 alleles (HLA A, B and DR) or 5 of 6 alleles, but not with mismatches at both alleles of a single locus (e.g. not mismatched for both HLA A alleles).
  Interventions: Biological: unrelated cord blood
- haplo BM with T cell depletion (Other): If there is no unrelated donor available meeting the matching criteria for unrelated bone marrow or unrelated cord blood donors.
  Interventions: Biological: haplo BM with T cell depletion
- unrelated PBSC with T cell depletion (Other): The preferred source will be bone marrow, however, if a donor is unable or unwilling to donate bone marrow, peripheral blood stem cells (PBSC) will be allowed.
  Interventions: Device: unrelated PBSC with T cell depletion

INTERVENTIONS:
Biological: unrelated BM with T cell depletion — Remaining unmanipulated bone marrow will be processed to isolate CD34+ cells (T cell depleted).
  Other Names: CD34+ selection using CliniMACS
  Arms: unrelated BM with T cell depletion
Biological: unrelated cord blood — Cord blood will be thawed (and processed if ABO incompatibility) per institutional SOP.
  Other Names: umbilical cord blood
  Arms: unrelated cord blood
Biological: haplo BM with T cell depletion — haplo-identical (parental) bone marrow will be processed for CD34+ cell isolation.
  Other Names: CD34+ selection with CliniMACS
  Arms: haplo BM with T cell depletion
Device: unrelated PBSC with T cell depletion — peripheral blood stem cell will be processed for CD34+ cell isolation.
  Other Names: CD34+ selection using CliniMACS
  Arms: unrelated PBSC with T cell depletion

SUMMARY:
This is a pilot clinical trial of hematopoietic stem cell transplantation for patients with a diagnosis of Severe Combined Immune Deficiency (SCID) who do not have an HLA-matched sibling donor. The stem cells will be derived from a 1) matched unrelated donor (MUD), 2) unrelated cord blood donor, or 3) a haplo-identical (parental) donor (in descending order of preference).Patients will receive a novel conditioning regimen with Busulfan, Fludarabine and Anti-thymocyte globulin (ATG) followed by an unrelated donor hematopoietic stem cell transplant (HSCT) with T-cell depletion using the CliniMACS device.

DETAILED DESCRIPTION:
The study is being conducted to assess the following:

* overall survival
* event-free survival (events are defined as: death,non-engraftment/2nd transplant, immune reconstitution failure)
* acute toxicity of the conditioning regimen
* engraftment frequency immune reconstitution frequency and tempo acute and chronic graft-versus-host disease (GVHD), frequency and severity.

The outcome from this protocol will be compared to the retrospective cohort consisting of all patients who have undergone haplo-identical HSCT for SCID at CHLA from 1984-2006 based on the assessment of the above-listed endpoints.

The CliniMACS device will be used for CD34+ selection in place of the Isolex 300i. The CliniMACS CD34 Reagent System is an investigational medical device that has not yet been approved by the FDA. This device is used in vitro to select and enrich specific cell populations. When using the CliniMACS CD34 Reagent, the system selects CD34+ cells from heterogenous hematological cell populations for transplantation in cases where this is clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* All patients with SCID who lack a histocompatible sibling or HLA-matched related donor will be considered as candidates for this study protocol.
* Eligible patients must have adequate physical function to tolerate the chemotherapy conditioning regimen and the HSCT, as measure by:

  1. Renal: creatinine clearance or GFR ≥50 ml/min/1.73m2, and not requiring dialysis
  2. Pulmonary: Because patients with SCID frequently present with infectious pneumonia causing ventilatory failure, patients will be considered for enrollment in the study even if respiratory failure requiring mechanical ventilatory support is present. In patients recently diagnosed with pneumonia, efforts to stabilize the respiratory status will be made prior to enrollment in the study.
  3. Infectious disease status. The presence of infection per se will not be a reason for exclusion from the study. Patients with SCID are frequently infected with both routine pathogens as well as opportunistic infections. Antibiotic, antifungal and antiviral prophylaxis and therapy will be instituted as clinically indicated. Despite the use of antimicrobial therapy, the ability to control infections will not be achieved unless HSCT is performed. Therefore, subjects may be enrolled in the study, even though infection is present, because control of infection may depend on engraftment of a donor immune system.
  4. Patients will be 0-21 years of age.

Exclusion Criteria:

* Patient with histocompatible sibling or other related donor
* End-organ failure that precludes the ability to tolerate the transplant procedure, including conditioning.
* Renal failure requiring dialysis
* Congenital heart disease resulting in congestive heart failure
* Severe CNS disease, e.g., coma or intractable seizures
* Ventilatory failure due to non-infectious etiology
* Major congenital anomalies that adversely affect survival, eg CNS malformations
* Metabolic diseases that would affect transplant survival, eg urea cycle disorders
* HIV infection

Since the only chance of survival for patients with SCID is successful transplantation, all patients with SCID will be considered to be potential subjects for the study, regardless of end-organ dysfunction.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2007-01-02 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neena Kapoor, M.D., Principal Investigator — Children's Hospital Los Angeles, University of Southern California
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unrelated BM With T Cell Depletion | Unrelated Cord Blood | Haplo BM With T Cell Depletion | Unrelated PBSC With T Cell Depletion
Started | 7 | 2 | 0 | 0
Completed | 6 | 1 | 0 | 0
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unrelated BM With T Cell Depletion | Unrelated Cord Blood | Haplo BM With T Cell Depletion | Unrelated PBSC With T Cell Depletion | Total
Number analyzed (Participants) | 7 | 2 | 0 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 2 | 0 | 0 | 9
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 |  |  | 1
  Male | 6 | 2 |  |  | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 0 | 5
  Not Hispanic or Latino | 3 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 1 | 0 |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 |  |  | 0
  White | 2 | 0 |  |  | 2
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 4 | 2 |  |  | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 |  |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Engraftment
Description: Engraftment is defined as recovery of blood counts (neutrophil and platelet engraftment) with cells of donor origin, documented by either bone marrow or peripheral blood chimerism assays after hematopoietic stem cell transplant.
Time Frame: 100 day
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated BM With T Cell Depletion | Unrelated Cord Blood | Haplo BM With T Cell Depletion | Unrelated PBSC With T Cell Depletion
Number analyzed (Participants) | 7 | 2 | 0 | 0
Participants | 7 | 2 |  |

2. Secondary Outcome: Number of Participants With Donor-derived CD3+ T Lymphocytes >/= 100/mm3
Description: Absolute number of donor-derived CD3+ T lymphocytes >/= 100/mm3 in participating subjects.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated BM With T Cell Depletion | Unrelated Cord Blood | Haplo BM With T Cell Depletion | Unrelated PBSC With T Cell Depletion
Number analyzed (Participants) | 7 | 2 | 0 | 0
Participants | 7 | 1 | 0 | 0

3. Other Pre Specified Outcome: Number of Participants With Veno-occlusive Disease (VOD) - Moderate and Severe
Description: Evaluation of veno-occlusive disease determined by the presence of the following features; fluid retention, weight gain, leaky capillary syndrome, painful liver enlargement, refractoriness to platelet tranfusion and hyperbilirubinemia
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated BM With T Cell Depletion | Unrelated Cord Blood | Haplo BM With T Cell Depletion | Unrelated PBSC With T Cell Depletion
Number analyzed (Participants) | 7 | 2 | 0 | 0
Participants | 2 | 1 | 0 | 0

4. Other Pre Specified Outcome: Number of Participants With Graft Versus Host Disease (GVHD) - Grade III or IV
Description: GVHD disease surveillance done by clinical evaluation, to include history, physical examination, specifically for rash, jaundice, liver dysfunction, nausea and vomiting, diarrhea and failure to thrive.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated BM With T Cell Depletion | Unrelated Cord Blood | Haplo BM With T Cell Depletion | Unrelated PBSC With T Cell Depletion
Number analyzed (Participants) | 7 | 2 | 0 | 0
Participants | 1 | 0 | 0 | 0

5. Other Pre Specified Outcome: Overall Survival
Description: Overalls survival of patient at 1 year post transplant
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Unrelated BM With T Cell Depletion | Unrelated Cord Blood | Haplo BM With T Cell Depletion | Unrelated PBSC With T Cell Depletion
Number analyzed (Participants) | 7 | 2 | 0 | 0
Participants | 6 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 1 year post transplant.
Arm/Group | Unrelated BM With T Cell Depletion | Unrelated Cord Blood | Haplo BM With T Cell Depletion | Unrelated PBSC With T Cell Depletion
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 5/7 | 1/2 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unrelated BM With T Cell Depletion (N=7) | Unrelated Cord Blood (N=2) | Haplo BM With T Cell Depletion (N=0) | Unrelated PBSC With T Cell Depletion (N=0)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Sinusoidal obstruction syndrome (SOS), previously known as veno-occlusive disease (VOD), is a distinctive and potentially fatal form of hepatic injury that occurs predominantly, if not only, after drug or toxin exposure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unrelated BM With T Cell Depletion (N=7) | Unrelated Cord Blood (N=2) | Haplo BM With T Cell Depletion (N=0) | Unrelated PBSC With T Cell Depletion (N=0)
Graft Versus Host Disease (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) — Graft versus host disease - condition post transplant the donor's immune cells in the transplant (graft) make antibodies against the patient's tissues (host) and attack vital organs (skin, GI track and liver common organs attacked)
Infection - Aspergillis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Pulmonary Aspergillis infection
Infection - Fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pulmonary fungal infection
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Busulfan toxicity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes